CLINICAL TRIAL: NCT01461707
Title: A Pilot Study of a Mobile Phone-Based Physical Activity Program in Pregnant Women
Brief Title: The MOTHER (Mobile Technologies to Help Enhancing Regular Physical Activity) Trial for Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 11-06992; 3R01HL104147-02S1 (NIH)
Record Dates: First submitted 2011-10-26; First posted 2011-10-28 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-10

CONDITIONS: Physical Activity
Keywords: Cellular phone; exercise; pregnant women; obesity; overweight; physical activity
MeSH Terms: conditions — Motor Activity; Obesity; Overweight | interventions — Fitness Trackers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mobile app plus activity monitor group (Experimental): Participants in the group will receive the mobile phone-based physical activity program and an activity monitor
  Interventions: Behavioral: Mobile phone-based physical activity; Behavioral: Activity monitor
- Activity monitor group (Active Comparator): Participants in the group will receive an activity monitor
  Interventions: Behavioral: Activity monitor

INTERVENTIONS:
Behavioral: Mobile phone-based physical activity — Participants will receive the mobile phone-based physical activity program using the trial app.
  Arms: Mobile app plus activity monitor group
Behavioral: Activity monitor — Participants will receive an activity monitor

SUMMARY:
Obesity among women of childbearing age and excessive weight gain during pregnancy are prevalent and steadily increasing health care issues. Regular physical activity is recommended to maintain healthy weight gain for pregnant women, however, a majority of pregnant women are sedentary. The investigators proposed to conduct a pilot study to estimate the potential efficacy of a mobile phone based physical activity intervention in 30 physically inactive pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* pregnant, gestational week (10-20 weeks)
* pre-pregnancy BMI ≥ 18.5 kg•m2
* physically inactive at work and during leisure time
* intent to be physically active
* access to a home telephone or a mobile phone
* have a personal computer access
* ability to communicate (speak and read) in English.

Exclusion Criteria:

* known medical or obstetric complication that restricts physical activity
* history of eating disorders
* current participation in lifestyle modification programs
* history of bariatric surgery.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-10; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JiWon Choi, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi J, Lee JH, Vittinghoff E, Fukuoka Y. mHealth Physical Activity Intervention: A Randomized Pilot Study in Physically Inactive Pregnant Women. Matern Child Health J. 2016 May;20(5):1091-101. doi: 10.1007/s10995-015-1895-7. PMID 26649879

RESULTS

PARTICIPANT FLOW:
Groups:
- Mobile App Plus Activity Monitor Group: Participants in the group will receive a study mobile phone application and an activity monitor
  Mobile phone-based physical activity program: Participants in the intervention group will receive an activity monitor and the mobile phone based physical activity intervention.
Period: Overall Study
Arm/Group | Mobile App Plus Activity Monitor Group | Activity Monitor Group
Started | 15 | 15
Completed | 14 | 15
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobile App Plus Activity Monitor Group | Activity Monitor Group | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.9 (2.5) | 34.5 (2.5) | 33.7 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 5 | 7 | 12
  Race: Black | 1 | 1 | 2
  Race: Hispanic/Latina | 2 | 1 | 3
  Race: White | 7 | 6 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Physical Activity Monitor Measured Steps
Description: Change in weekly mean steps per day
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: step
Arm/Group | Mobile App Plus Activity Monitor Group | Activity Monitor Group
Number analyzed (Participants) | 14 | 15
step
  Baseline to week 1-4 | 1166.6 (1709.4) | 1062.6 (2325.5)
  Baseline to week 5-8 | 1092.1 (1925.3) | 804.3 (1752.9)
  Baseline to week 9-12 | 1096.2 (1898.1) | 258.7 (1603.7)

2. Secondary Outcome: 7-Day Physical Activity Recall
Description: Change in mean energy expenditure
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Mobile App Plus Activity Monitor Group | Activity Monitor Group
Number analyzed (Participants) | 14 | 15
kcal/day | 69 (223.1) | 204.3 (314.7)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Mobile App Plus Activity Monitor Group | Activity Monitor Group
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No